CLINICAL TRIAL: NCT05548296
Title: A Phase 2 Study of ACR-368 Therapy in Subjects With Endometrial Cancer
Brief Title: A Phase 2 Study of ACR-368 in Endometrial Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acrivon Therapeutics (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACR-368-201 (GOG 3082)
Record Dates: First submitted 2022-08-29; First posted 2022-09-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Adenocarcinoma
Keywords: Endometrial Cancer; Endometrial Neoplasm; Ultralow dose gemcitabine; ACR-368
MeSH Terms: conditions — Endometrial Neoplasms | interventions — prexasertib; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Participants with an OncoSignature Positive test will enter the Arm 1 cohort that will assess the efficacy of ACR-368 as monotherapy in endometrial cancer. Participants with an OncoSignature Negative test will enter the Arm 2 cohort to assess the efficacy and safety of ACR-368 with ULDG sensitization. Participants without OncoSignature testing will enter an OncoSignature Unselected Arm 3 cohort to assess the efficacy and safety of ACR-368 with ULDG sensitization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- OncoSignature Positive Tumors (Experimental): ARM 1: Participants with OncoSignature Positive Tumors will enter a Phase 2 Simon 2-Stage Study that will assess the efficacy of ACR-368 as monotherapy.
  Interventions: Drug: ACR-368; Diagnostic Test: OncoSignature
- OncoSignature Negative Tumors (Experimental): Arm 2: Participants with OncoSignature Negative Tumors will receive ACR-368 with ULDG sensitization. The Phase 2 Study will assess the efficacy and safety of ACR-368 with ULDG sensitization.
  Interventions: Drug: ACR-368; Drug: Gemcitabine; Diagnostic Test: OncoSignature
- OncoSignature Unselected (All-Comers) (Experimental): Arm 3: Participants who are OncoSignature Unselected will receive ACR-368 with ULDG sensitization. The Phase 2 Study will assess the efficacy and safety of ACR-368 with ULDG sensitization.
  Interventions: Drug: ACR-368; Drug: Gemcitabine

INTERVENTIONS:
Drug: ACR-368 — ACR-368 is an experimental drug
  Other Names: prexasertib
Drug: Gemcitabine — Sensitization of tumor cells is provided through administration of ULDG
  Arms: OncoSignature Negative Tumors; OncoSignature Unselected (All-Comers)
Diagnostic Test: OncoSignature — Prospective prediction of drug sensitivity based on a pretreatment tumor biopsy
  Arms: OncoSignature Negative Tumors; OncoSignature Positive Tumors

SUMMARY:
This is an open label Phase 2 study to evaluate the efficacy and safety of ACR-368 as monotherapy or with ultra-low dose gemcitabine (ULDG) sensitization in participants with endometrial cancer.

DETAILED DESCRIPTION:
OncoSignature Selected Cohorts (Arms 1 and 2):

Participants in Arms 1 & 2 will be allocated into two arms based on prospectively predicted sensitivity to ACR-368 using the OncoSignature® Companion Diagnostic test, as follows:

Arm 1: OncoSignature Positive tumors

Arm 2: OncoSignature Negative tumors

OncoSignature Unselected Cohort (Arm 3):

In Arm 3 participants will not require a biopsy or OncoSignature result.

Participants in Arm 1 will receive ACR-368 as monotherapy. Participants in Arms 2 and 3 will receive ACR-368 with ULDG sensitization. Participants in all arms will be treated until disease progression, unacceptable toxicity or any criterion for stopping the study drug or withdrawal from the trial occurs.

Arms 1 and 2 do not apply to sites in the European Union (EU), which will enroll subjects in Arm 3.

ELIGIBILITY:
Inclusion Criteria: General

1. Participant must be able to give signed, written informed consent.
2. Participant must have histologically documented, high-grade endometrial cancer. Arms 1 and 2

   1. All high-grade epithelial endometrial histological subtypes are eligible including: endometrioid (Grade 3 only), serous, carcinosarcomas, clear-cell carcinoma, and mixed histologies.

      Arm 3
   2. Serous carcinoma or mixed tumors with a majority component of serous carcinoma or carcinosarcoma where the carcinomatous component is serous carcinoma.
3. Treatment History Requirements:

   Arms 1 and 2
   1. Subject must have received prior platinum-based chemotherapy
   2. Subject must have received prior anti-PD-(L)1 therapy
   3. Subject must not have received more than three lines of prior systemic therapy Arm 3

   <!-- -->

   1. Subject must have received prior platinum-based chemotherapy
   2. Subject must have received prior anti-PD-(L)1 therapy
   3. Subject must not have received more than two lines of prior systemic therapy
4. Participant must have histologically confirmed metastatic cancer that has progressed during or after at least 1 prior therapeutic regimen.
5. Participant must have at least 1 measurable lesion per RECIST v1.1 criteria (by local Investigator) in a baseline tumor imaging that has been obtained within 28 days of the treatment start. Participant must have radiographic evidence of disease progression based on RECIST v1.1 criteria following the most recent line of treatment.
6. Arm 1 and 2 only: Participant must be willing to provide tissue from a newly obtained tumor biopsy from an accessible tumor lesion not previously irradiated after written informed consent.

   Newly obtained is defined as a specimen taken after written informed consent is obtained, during the 28-day Screening period.

   Note: Subjects at EU sites are not eligible for Arm 1 and Arm 2
7. Participant must be willing to provide an archival tumor tissue block or at least 20 unstained slides, if available.
8. Participant must have stabilized or recovered (Grade 1 or baseline) from all prior therapy related toxicities, except as follows:

   1. Alopecia is accepted.
   2. Endocrine events from prior immunotherapy stabilized at ≤ Grade 2 due to need for replacement therapy are accepted (including hypothyroidism, diabetes mellitus, or adrenal insufficiency).
   3. Neuropathy events from prior cytotoxic therapies stabilized at ≤ Grade 2 are accepted.
9. Participant must have an Eastern Cooperative Oncology Group Performance Status 0 or 1.
10. Participant must have an estimated life expectancy of longer than 3 months.
11. Participant must have adequate organ function at Screening, defined as:

    1. Absolute neutrophil count > 1500 cells/µL without growth factor support within 1 week prior to obtaining the hematology values at Screening.
    2. Hemoglobin ≥ 9.0 g/dL.
    3. Platelets ≥ 150,000 cells/µL without transfusion within 1 week prior to obtaining the hematology values at Screening.
    4. Renal function is defined as Glomerular filtration rate (GFR) ≥ 50 mL/min/1.73m2. Note: GFR may be estimated using site standard methods (e.g., CKD-EPI, MDRD, or Cockcroft-Gault) or measured using 24-hour urine collection or Chrome-EDTA clearance, as per site standard practice.
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); ≤ 5 × ULN if liver metastases are present.
    6. Total bilirubin ≤ 1.5 × ULN not associated with Gilbert's syndrome. If associated with Gilbert's syndrome ≤ 3 x ULN is acceptable.
    7. Serum albumin ≥ 3 g/dL.
12. Participant must have adequate coagulation profile as defined below if not on anticoagulation. If subject is receiving anticoagulation therapy, then subject must be on a stable dose of anticoagulation for ≥ 1 month:

    1. Prothrombin time within 1.5 x ULN.
    2. Activated partial thromboplastin time within 1.5 x ULN.

Exclusion Criteria: General

1. Participant with known symptomatic brain metastases requiring > 10 mg/day of prednisolone (or its equivalent). Participants with previously diagnosed brain metastases are eligible if they have completed their treatment, have recovered from the acute effects of radiation therapy or surgery prior to the start of ACR-368 treatment, fulfill the steroid requirement for these metastases, and are neurologically stable based on central nervous system imaging ≥ 4 weeks after treatment.
2. Participant has mesenchymal tumors of the uterus.
3. Participant has a history of clinically meaningful ascites, defined as history of paracentesis or thoracentesis with therapeutic intent, within 4 weeks of Screening. Subjects with planned therapeutic paracentesis or thoracentesis between Screening and Cycle 1 Day 1 dosing are excluded.
4. Participant had systemic therapy or radiation therapy within 3 weeks prior to the first dose of study drug.
5. Participants has known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection that is considered uncontrolled based on the criteria included in Appendix 2.
6. Participant has a history of clinically meaningful coagulopathy, bleeding diathesis.
7. Participant has cardiovascular disease, defined as:

   1. Uncontrolled hypertension defined as blood pressure > 160/90 mmHg at Screening confirmed by repeat (medication permitted).
   2. History of torsades de pointes, significant Screening electrocardiogram (ECG) abnormalities, including ventricular rhythm disturbances, unstable cardiac arrhythmia requiring medication, pathologic symptomatic bradycardia, left bundle branch block, second degree atrioventricular (AV) block type II, third degree AV block, Grade ≥ 2 bradycardia, uncorrected hypokalemia not amenable to correction, congenital long QT syndrome, prolonged QT interval due to medications, corrected QT based on Fridericia's formula (QTcF) > 450 msec (for men) or > 470 msec (for women).
   3. Symptomatic heart failure (per New York Heart Association guidelines; (Caraballo, 2019), unstable angina, myocardial infarction, severe cardiovascular disease (ejection fraction < 20%, transient ischemic attack, or cerebrovascular accident within 6 months of Day 1).
8. Participant has a history of major surgery within 4 weeks of Screening.
9. Participant has experienced bowel obstruction related to the current cancer within the last 6 months or signs or symptoms of intestinal obstruction, which include nausea, vomiting, or objective radiologic finding of bowel obstruction in the last 4 weeks before the start of the treatment.
10. Participant has taken a prior cell cycle CHK1 inhibitor, including ACR-368

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Arm 1: Anti-tumor activity of ACR-368 in Endometrial cancer subjects that are OncoSignature Positive. | Response will be assessed every 8 weeks from baseline through 2 years or death.
  Assess Objective Response Rate (ORR) per RECIST v1.1 by computed tomography or magnetic resonance imaging.
Arm 2: Anti-tumor activity of ACR-368 with ULDG sensitization in Endometrial cancer subjects that are OncoSignature Negative. | Response will be assessed every 8 weeks from baseline through 2 years or death.
  Objective Response Rate (ORR) per RECIST v1.1 by computed tomography or magnetic resonance imaging.
Arm 3: Anti-tumor activity of ACR-368 with ULDG sensitization in Endometrial cancer subjects (All-Comers). | Response will be assessed every 8 weeks from baseline through 2 years or death.
  Objective Response Rate (ORR) per RECIST v1.1 by computed tomography or magnetic resonance imaging.

SECONDARY OUTCOMES:
Arm 1: Adverse Events (AEs) for ACR-368 | AEs will be assessed from baseline through 2 years or death.
  Safety will be assessed by the incidence of AEs characterized overall and by type, incidence, severity graded according to NCI CTCAE v5.0, seriousness, and relationship to study treatment.
Arm 2 and Arm 3: Adverse Events (AEs) for ACR-368 with ULDG sensitization | AEs will be assessed from baseline through 2 years or death.
  Safety will be assessed by the incidence of AEs characterized overall and by type, incidence, severity graded according to NCI CTCAE v5.0, seriousness, and relationship to study treatment.
All Arms: Limited pharmacokinetic (PK) testing. | Dose of ACR-368 at day 1 and day 15 of first cycle.
  Cmax and Tmax will be assessed in the first cycle. Blood samples will be collected at baseline, end of infusion, hour 2 and hour 4.
Overall Survival (OS) | Up to 2 years
  The time from date of enrollment until date of death.
Duration of Response (DOR) | Up to 2 years
  The time from initial response until investigator assessed progressive disease for all subjects who achieve a confirmed objective response.
Progression-free Survival (PFS) | Up to 2 years
  The time from date of enrollment until disease progression or death whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, Principal Investigator — Dana-Farber Cancer Institute (DFCI); Isabelle Ray-Coquard, MD, Principal Investigator — Centre Leon Berard
Locations (90):
- United States (69):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Center, Anchorage, Alaska
  - HonorHealth, Phoenix, Arizona
  - Arizona Oncology Associate, PC- HOPE, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Cancer Center, Newport Beach, California
  - UC Irvine Health, Orange, California
  - Stanford Cancer Center, Palo Alto, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Gynecologic Oncology/Regional Cancer Center, Fort Myers, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Ascension St. Vicent Hospital, Inc., Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - LSU Health Sciences, New Orleans, Louisiana
  - Trials365, LLC, Shreveport, Louisiana
  - American Oncology Partners of Maryland PA, Bethesda, Maryland
  - National Institutes of Health, Clinical Center, Bethesda, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - HCA Midwest, Kansas City, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai Health System, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Hilliard, Ohio
  - Stephenson Cancer Center at OU Health, Oklahoma City, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Oregon Health & Sciences University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Sanford Health, Sioux Falls, South Dakota
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Summit Cancer Center, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- France (4):
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Insitute de Cancérologie de l'Ouest, Saint-Herblain
  - Institute Gustave Roussy, Villejuif
- Germany (3):
  - KEM | Evang. Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Münster, Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - Universitätsklinikum Ulm, Frauenheilunde und Geburtshilfe, Ulm
- Italy (7):
  - CRO Aviano, Aviano
  - Istituto Clinico Cannizzaro Catania, Catania
  - Istituto Europeo di Oncologia, Milan
  - Fondazione Pascale Istituto Tumori, Napoli
  - Humanitas University, Pieve Emanuele
  - Policlinico Gemelli, Roma
  - Ospedale Mauriziano Torino, Turin
- Spain (7):
  - Hospital Clínic de Barcelona, Barcelona
  - Institut Català of Oncology (ICO), Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://acrivon.com